CLINICAL TRIAL: NCT00382694
Title: Fludarabine Added to Induction Treatment in Untreated Multiple Myeloma Patients: A Randomised, Placebo Controlled, Double Blind Phase II Trial: NMSG #13/03
Brief Title: Fludarabine Added to Induction Treatment in Untreated Multiple Myeloma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nordic Myeloma Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMSG#13/03
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2006-09-29 (Estimated); Status verified 2006-09

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Induction therapy; High-dose melphalan; Autologous stem cell support; Fludarabine; Cyclophosphamide; Dexamethasone; Safety; Toxicity
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — fludarabine

INTERVENTIONS:
Drug: Fludarabine

SUMMARY:
Multiple myeloma is an incurable malignant disease which evnetuelly will relapse after primary treatment. Clonal B-cells have been identified and in theory these cells might be sleeping during primary treatment and be responsible for later relapse. Fluarabine has documented effect on both resting and dividing cells including B-cells. The protocol aim at evaluating safety and toxicity of adding fludarabine to induction chemotherapy with cyclophosphamide and dexamethasone before high-dose melphalan with autologous stem cell support.

DETAILED DESCRIPTION:
This is a randomised, placebo controlled, phase II study evaluating toxicity and safety of fludarabine added to CyDex (cyclophosphamide+dexamethasone) as induction therapy in younger patients with untreated and treatment demanding multiple myeloma. The treatment regimen Patients will be randomised at diagnosis either to CyDex + Placebo (control Arm A) or CyDex + Fludarabine (Experimental Arm B).

OBJECTIVES:

* Primary:To determine the toxicity and safety of fludarabine when added to induction therapy by registration of side effects and adverse events in accordance with the common toxicity criteria (CTC).
* Secondary:To quantitate clonal cells in bone marrow and blood by flow cytometry (MRD)and to study new potential prognostic markers identified by cytomic, genomic and proteomic analysis.
* Tertiary: To estimate the efficacy of fludarabine when added to induction chemotherapy(CyDex) in patients with multiple myeloma by clinical end points: disease response and progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma, stage I-III, previously untreated, and eligible for induction therapy followed by high dose treatment supported by autologous stem cell transplantation.

Exclusion Criteria:

* Severe uncontrolled clinical or microbiological evidence of infection at the time of enrolment.
* Other active malignancy.
* Severe coincident heart or lung disease including uncontrolled hypertension, unstable angina, congestive heart failure, coronary angioplasty within six months, myocardial infarction within the last six months, or uncontrolled cardiac arrhythmia.
* Other severe illness including poorly controlled diabetes.
* Haemolytic anaemia (Coombs positive without evidence of haemolysis is accepted).
* Idiopathic thrombocytopenic purpura.
* Terminal illness.
* Allogenic transplantation planned within 6 months.
* Chemotherapy before inclusion.
* Pregnancy or breast-feeding, or inadequate contraceptive precautions.
* Psychiatric disease, abuse of alcohol or narcotics, or any other disorder that might compromise the patients ability to give informed consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80
Dates: Start 2005-05; Study Completion 2006-12

PRIMARY OUTCOMES:
The toxicity and safety of Fludarabine when added to induction therapy by registration of side effects and adverse events in accordance with the common toxicity criteria (CTC).

SECONDARY OUTCOMES:
Quantification of clonal cells in bone marrow and blood by flow cytometry (MRD) and to study new potential prognostic markers identified by cytomic, genomic and proteomic analysis.
Estimation of the efficacy of Fludarabine when added to induction chemotherapy (CyDex) in patients with multiple myeloma by clinical end points: disease response and progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Hans E. Johnsen, Prof., MD, Principal Investigator — Aalborg Univeristy Hospital
Locations (6):
- Denmark (6):
  - Department of Haematology B, Aalborg Hospital, University of Aarhus, Aalborg
  - Dept. of Haematology, Århus University Hospital, Aarhus
  - Department of Haematology, Herlev University Hospital, Herlev
  - Department of Haematology, Rigshospitalet, København Ø
  - Department of Haematology X, Odense University Hospital, Odense
  - Department of Haematology, Vejle Hospital, Vejle